CLINICAL TRIAL: NCT01887080
Title: Effects of Microcurrent in a Cardiovascular Rehabilitation Home-based Program in Patients With Acute Myocardial Infarction
Brief Title: Effects of Microcurrent in a Cardiovascular Rehabilitation Home-based Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Superior de Tecnologia da Saúde do Porto (Other)
Responsible Party: Principal Investigator, Andreia Noites, Professor, Escola Superior de Tecnologia da Saúde do Porto
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: AN-002
Record Dates: First submitted 2013-06-18; First posted 2013-06-26 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2014-01

CONDITIONS: Acute Myocardial Infarction
Keywords: Cardiovascular rehabilitation home-based; Acute myocardial infarction; Obesity; Microcurrent
MeSH Terms: conditions — Obesity | interventions — Exercise; Heart Disease Risk Factors

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Exercise (Experimental): Experimental group 1 performed cardiovascular rehabilitation home-based program
  Interventions: Other: Exercise; Other: Cardiovascular Risk Factors
- Exercise afther Microcurrent (Experimental): Experimental group 2 performed cardiovascular rehabilitation home-based program just after microcurrent.
  Interventions: Other: Exercise; Device: Microcurrent; Other: Cardiovascular Risk Factors
- Cardiovascular Risk Factors (Other): Education about risk factors
  Interventions: Other: Cardiovascular Risk Factors

INTERVENTIONS:
Other: Exercise — This group had the exercise program, thrice a week for eight weeks.
  The exercise protocol consists of 10 exercises: aerobic and resistance exercises. It was used a moderate intensity (60% of maximum heart rate of stress test with progression until 80%). Subjects were taught to monitor exercise intensity by measuring the manual heart rate, by using the scale of perceived exertion Borg (11-13), and by observation of signs.
  The exercise protocol was done with supervision from a distance, using information technologies (SMS, phone, email ...), and when necessary it was resorted to routine meetings.
  Arms: Exercise; Exercise afther Microcurrent
Device: Microcurrent — This group had the exercise program after electrolipolysis, thrice a week for eight weeks.
  The electrolipolysis consisted of 30-minute sessions: the first 15 minutes with a frequency of 30 Hz and the final 15 minutes with a frequency of 10 Hz; with a pulse time of 10 ms; and an intensity below the threshold of sensitivity (with a maximum of 750 μA). There were used 4 transcutaneous electrodes in the abdominal region (parallel position).
  Microcurrent was done with supervision from a distance, using information technologies (SMS, phone, email ...), and when necessary it was resorted to routine meetings.
  Arms: Exercise afther Microcurrent
Other: Cardiovascular Risk Factors — It was handed flyers on major cardiovascular risk factors: cholesterol, obesity, diabetes, smoking and hypertension.

SUMMARY:
The aim of this study was to investigate the effects of electric stimulation (electrolipolysis) in a home-based cardiovascular rehabilitation program in patients with acute myocardial infarction

DETAILED DESCRIPTION:
Cardiovascular disease is the leading cause of death in most industrialized countries.

It is widely accepted that cardiac rehabilitation has a beneficial role in the control of modifiable cardiovascular risk factors. However, these cardiovascular rehabilitation programs are scarce and only a small fraction of the population who needs has access. So, it is pertinent to the displacement of these programs to the community context.

Obesity has become a truly global epidemic among children and adults, as well as changing the metabolic profile: when occurs an excessive accumulation of adipose tissue (mainly central distribution) there are a set of changes / adjustments to the cardiac structure and function. The electrical stimulation of abdominal subcutaneous (electrolipolysis) is a procedure often used in physical therapy clinics to reduce waist circumference. However, the effectiveness of this intervention, the selection of parameters, and the duration of its effects in cardiac patients are not yet clarified in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Individuals admitted to the coronary care unit for acute myocardial infarction for more than one year;
* Individuals of both sexes;
* Ages between 40 and 75 years;
* Heart disease stabilized;
* Motivation to perform physical activity for 8 weeks;
* Cognitive level sufficient to understand the particulars of the study.

Exclusion Criteria:

* Contraindications of micro-current (pacemaker, osteosynthesis material, tumor areas and open wounds or skin changes in the abdominal region);
* Pregnant at the time, in the preceding 6 months or wishing to become pregnant during the intervention period;
* Neurological, musculoskeletal or respiratory disorders;
* Individuals who are to carry out other therapies.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-09; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory Fitness | Change from Baseline in Cardiorespiratory Fitness at 8 weeks of Cardiac Rehabilitation Home-based Program
  The stress test was performed according to the Bruce protocol on a treadmill. The test begins with the treadmill set to a low speed (2.7 km/h) and a 10% incline, and every 3 minutes the speed and angle of incline are increased. Generally the incline is increased by 2% at every level, until exhaustion.
  It was measured resting, maximum and recovery heart rate; resting, maximum and recovery systolic blood pressure; resting, maximum and recovery diastolic blood pressure; resting, maximum and recovery double product; time and recovery time; speed; slope; and changes in functional capacity.
Blood tests | Change from Baseline in blood tests at 8 weeks of Cardiac Rehabilitation Home-based Program
  They were performed in the morning after fasting for about 12 hours, to avoid the interference of postprandial lipemia.
  It was measured glucose, cholesterol and triglycerides.
Computerized axial tomography | Change from Baseline in Computerized axial tomography at 8 weeks of Cardiac Rehabilitation Home-based Program
  It was measured subcutaneous, visceral and total abdominal fat.

SECONDARY OUTCOMES:
Bioimpedance values | Change from Baseline in Bioimpedance values at 8 weeks of Cardiac Rehabilitation Home-Based Program and 4 Weeks After Finishing the Protocol
  I twas used a bioimpedance scale (BIO) InnerScan Tanita, TBF-300A, which uses four electrodes (two on each foot) for the passage of an electric current. People were told to undress her clothes and stay only shorts without metal objects.
Perimeters measurements | Change from Baseline in Perimeters measurements at 8 weeks of Cardiac Rehabilitation Home-based Program and 4 Weeks After Finishing the Protocol
  The perimeters measurements were done, at the end of expiration, at waist level (below last rib), at navel level, at the point immediately above the iliac crests and at trochanters level. The waist-hip ratio was calculated using the waist level perimeter divided by trochanters level perimeter
Skinfolds measurements | Change from Baseline in Skinfolds measurements at 8 weeks of Cardiac Rehabilitation Home-based Program and 4 Weeks After Finishing the Protocol
  Subscapular, Triceps, Biceps, Suprailiac, vertical and horizontal abdominal skinfolds were performed three times in right hemi body, by Harpenden Caliper
Daily Physical Activity | Change from Baseline in Daily Physical Activity at 8 weeks of Cardiac Rehabilitation Home-based Program and 4 Weeks After Finishing the Protocol
  Physical activity will be objectively measured for 7 consecutive days using the ActiGraph accelerometer (model GT3X, Florida, USA).
Flexicurve spinal measurement | Change from Baseline in Flexicurve Spinal Measurement at 8 weeks of Cardiac Rehabilitation Home-based Program and 4 Weeks After Finishing the Protocol
  It was proceeded 3 measurements with flexicurve, with references of C7 and L1 to calculate the thoracic index.
Y-Balance Test | Change from Baseline in Y-Balance Test at 8 weeks of Cardiac Rehabilitation Home-based Program and 4 Weeks After Finishing the Protocol at 8 weeks of Cardiac Rehabilitation Home-based Program and 4 Weeks After Finishing the Protocol
  The Y-balance test assesses anterior, posteromedial and posterolateral components.
One Leg Standing Test | Change from Baseline in One Leg Standing Test at 8 weeks of Cardiac Rehabilitation Home-based Program and 4 Weeks After Finishing the Protocol
  It was recorded the best time, for two lower extremities (until the maximum of 30 seconds), without unbalancing . It was made with the eye open and closed.

OTHER OUTCOMES:
Food Frequency Questionnaire | Change from Baseline in Food Frequency Questionnaire at 8 weeks of Cardiac Rehabilitation Home-based Program and 4 Weeks After Finishing the Protocol
  Food Frequency Questionnaire was used to monitor lifestyle during sessions.
International Physical Activity Questionnaire | Change from Baseline in International Physical Activity Questionnaire at 8 weeks of Cardiac Rehabilitation Home-based Program and 4 Weeks After Finishing the Protocol
  Moderate physical activity level was used to monitor lifestyle during sessions
Depression Anxiety Stress Scales (DASS-21) | Change from Baseline in DASS-21 at 8 weeks of Cardiac Rehabilitation Home-based Program and 4 Weeks After Finishing the Protocol
  Depression Anxiety Stress Scales was used to monitor lifestyle during sessions
MacNew Heart Disease health-related quality of life instrument | Change from Baseline in MacNew at 8 weeks of Cardiac Rehabilitation Home-based Program and 4 Weeks After Finishing the Protocol
  MacNew was used to monitor lifestyle during sessions
EuroQoL Quality of Life Scale (EQ-5D) | Change from Baseline in EQ-5D at 8 weeks of Cardiac Rehabilitation Home-based Program and 4 Weeks After Finishing the Protocol
  EQ-5D was used to monitor lifestyle during sessions
Montreal Cognitive Assessment(MOCA) | Change from Baseline in MOCA at 8 weeks of Cardiac Rehabilitation Home-based Program and 4 Weeks After Finishing the Protocol
  Moca was used to monitor lifestyle during sessions
Transtheoretical Model Exercise Behavior | Change from Baseline in Transtheoretical Model Exercise Behavior at 8 weeks of Cardiac Rehabilitation Home-based Program and 4 Weeks After Finishing the Protocol
  Transtheoretical Model Exercise Behavior consists of four subscales:
  1. Identify the stages of exercise behavior
  2. Processes of change of exercise behavior
  3. Decisional balance of exercise behavior
  4. Self-efficacy of exercise behavior

CONTACTS AND LOCATIONS:
Overall Officials: Andreia Noites, MSc, Principal Investigator — Escola Superior de Tecnologia da Saúde do Porto; Carla Patricia Freitas, MSc, Principal Investigator — Escola Superior de Tecnologia da Saúde do Porto; Joana Moura Pinto, MSc, Principal Investigator — Escola Superior de Tecnologia da Saúde do Porto
Locations (1):
- Andreia Noites, Porto, Vila Nova de Gaia, Portugal

REFERENCES:
- [Result] Williams MA, Haskell WL, Ades PA, Amsterdam EA, Bittner V, Franklin BA, Gulanick M, Laing ST, Stewart KJ; American Heart Association Council on Clinical Cardiology; American Heart Association Council on Nutrition, Physical Activity, and Metabolism. Resistance exercise in individuals with and without cardiovascular disease: 2007 update: a scientific statement from the American Heart Association Council on Clinical Cardiology and Council on Nutrition, Physical Activity, and Metabolism. Circulation. 2007 Jul 31;116(5):572-84. doi: 10.1161/CIRCULATIONAHA.107.185214. Epub 2007 Jul 16. PMID 17638929
- [Result] Hamida ZH, Comtois AS, Portmann M, Boucher JP, Savard R. Effect of electrical stimulation on lipolysis of human white adipocytes. Appl Physiol Nutr Metab. 2011 Apr;36(2):271-5. doi: 10.1139/h11-011. PMID 21609289
- [Result] Donnelly JE, Blair SN, Jakicic JM, Manore MM, Rankin JW, Smith BK; American College of Sports Medicine. American College of Sports Medicine Position Stand. Appropriate physical activity intervention strategies for weight loss and prevention of weight regain for adults. Med Sci Sports Exerc. 2009 Feb;41(2):459-71. doi: 10.1249/MSS.0b013e3181949333. PMID 19127177
- [Derived] Noites A, Freitas CP, Pinto J, Melo C, Vieira A, Albuquerque A, Teixeira M, Ribeiro F, Bastos JM. Effects of a Phase IV Home-Based Cardiac Rehabilitation Program on Cardiorespiratory Fitness and Physical Activity. Heart Lung Circ. 2017 May;26(5):455-462. doi: 10.1016/j.hlc.2016.08.004. Epub 2016 Sep 13. PMID 27743855